CLINICAL TRIAL: NCT02307474
Title: CASE 10813: A Pilot Study of SBRT With Adjuvant Pazopanib for Renal Cell Carcinoma
Brief Title: A Pilot Study of SBRT With Adjuvant Pazopanib for Renal Cell Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE10813; NCI-2014-02275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE10813 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma
Keywords: Kidney; Renal Cell Carcinoma; Cancer; Pilot; Pazopanib; stereotactic body radiation therapy; SBRT
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Radiosurgery; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Stereotactic Radiosurgery, pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO daily for up to 60 days. Patients then continue to receive pazopanib hydrochloride PO daily and undergo stereotactic radiosurgery (SBRT) every other day over days 60-65.
  Interventions: Radiation: Stereotactic Radiosurgery; Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — 3 fractions of 16 Gy per fraction to a total dose of 48 Gy on non-consecutive day within a 10 day time span
  Other Names: SBRT; Stereotactic External Beam Irradiation; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; Stereotactic Body Radiation Therapy
Drug: Pazopanib Hydrochloride — Given PO starting at 800mg to be systematically altered following drug related toxicities.
  Other Names: GW786034B; Votrient; pazopanib

SUMMARY:
This pilot clinical trial studies the side effects of stereotactic body radiation therapy and pazopanib hydrochloride in treating patients with kidney cancer who are not able to undergo surgery. Stereotactic body radiation therapy is a specialized radiation therapy that delivers high doses of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Pazopanib hydrochloride may stop the growth of tumor cells by blocking an enzyme needed for cell growth. Giving pazopanib hydrochloride before stereotactic body radiation therapy may help make the tumor smaller and be an alternative treatment for patients who cannot undergo surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of treatment related toxicity reports following stereotactic body radiation therapy (SBRT) and pazopanib (pazopanib hydrochloride) as a determination of the tolerability of combined therapy in patients with clear cell renal cell carcinoma (RCC).

SECONDARY OBJECTIVES:

I. To determine the tumor diameter/volume change prior to and following pazopanib treatment prior to SBRT.

II. To determine the impact of pre SBRT pazopanib therapy on radiation therapy target volumes for evidence of tumor shrinkage.

III. To evaluate tumor change in radiation therapy target volumes and the incidence of treatment related toxicity reports and sparing of non-involved nephron.

IV. Report change in tumor control following pazopanib and SBRT as evaluated by post treatment repeat biopsy and/or Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) daily for up to 60 days. Patients then continue to receive pazopanib hydrochloride PO daily and undergo SBRT every other day over days 60-65.

After completion of study treatment, patients are followed up at 1, 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is considered a poor surgical candidate for removal of a renal mass as determined by pre-operative assessment due to the following factors or various combinations thereof:

  * Significant comorbidity precluding ability to deliver anesthesia, without compromised ability to undergo systemic chemotherapy with pazopanib as deemed by the Urologist and Medical Oncologist
  * Medically documented contraindication for surgery due to religion or risk of blood transfusion
  * Size or location of tumor deemed high risk for surgical intervention by Urologist
  * Unacceptable risk for anesthesia, such as history of malignant hyperthermia
  * Any one of these factors may or may not constitute unresectability, but for consideration for this trial, the surgical and medical oncologist must agree that the particular constellation of findings for the patient under consideration would likely entail a low probability (< 50%) that the tumor would be resectable (with negative margins) or that the potential morbidity associated with an attempt at surgical resection would not be clinically acceptable
  * The numerical thresholds noted above are only a guideline and the clinical judgment of the surgeon and medical oncologist will determine unresectability or if patient refuses surgery or other forms of local therapy; the histopathology for this cohort is limited to clear cell carcinoma of the kidney
* Patient is able to give and sign study specific informed consent
* Negative serum or urine pregnancy test within 72 hours prior to registration for women of childbearing potential and agrees to use contraception for the duration of the treatment cycle and for a minimum of 30-days following the end of therapy (a minimum estimate 95 days)
* Patient has a pathologically confirmed diagnosis of clear cell RCC
* Karnofsky status of ≥ 70%
* Subject has no contraindication for computed tomography (CT) and/or magnetic resonance imaging (MRI) during screening and is able to complete a screening examination; CT and/or MRI within 6 months of screening is required
* Patient has inadequate organ function as defined by:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x laboratory upper limit of normal (ULN)
  * Total serum bilirubin < 1.5 x ULN
  * Absolute neutrophil count (ANC) > 1500/uL
  * Platelets > 100,000/uL
  * Hemoglobin > 9.0 g/dL (no transfusion permitted within 1 week)
  * Serum creatinine < 2.5 mg/dL
  * Urine to protein to creatinine (UPC) ratio < 1; if UPC > 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible
  * Prothrombin time (PT) or international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.2 X upper limit of normal (ULN)

Exclusion Criteria:

* Any patient with active connective tissue disease such as lupus, dermatomyositis
* Major psychiatric illness, which would prevent completion of treatment or interfere with follow-up
* Prior dose of radiation overlapping the treatment field determined by a study Radiation Oncologist to represent unacceptable risk for additional radiation to be targeted to the field
* Pregnant and lactating females, and unwillingness to use contraception; or male subject not willing to use contraception during and for 21 days after the last dose of pazopanib therapy
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding (e.g. active peptic ulcer, ulcerative colitis, Crohn's disease, abdominal fistula) within prior 6 months
* Clinically significant gastrointestinal abnormalities that may affect absorption (e.g. malabsorption syndrome, major resection of the stomach or small bowel)
* Corrected QT interval (QTc) > 480 msecs (record QTc correction method)
* History of clinically significant cardiovascular condition with the past 6 months (e.g. angioplasty or stenting, myocardial infarction, unstable angina, bypass surgery, symptomatic peripheral arterial disease [PAD], class III or IV congestive heart failure)
* History of cerebrovascular accident within the past 6 months (e.g. transient ischemic attack [TIA])
* Poorly controlled hypertension (systolic blood pressure [SBP] >= 140 mmHg or diastolic blood pressure [DBP] >= 90 mmHg); the initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry
* Major surgery or trauma within 29 days prior to first dose of study drug and/or presence of any non-healing wound, fracture or ulcer (catheter placement is not major surgery)
* Evidence of active bleeding or bleeding diathesis
* Recent hemoptysis (>= half teaspoon of red blood within 8 weeks before first dose of study drug)
* Treatment with any other anti-cancer therapies (e.g. other radiation, surgery or tumor embolization) within the last 14 days prior to first dose of study drug; or chemotherapy, immunotherapy, biologic therapy, investigational or hormonal therapy within 14-days (or 5 half-lives of a drug whichever is longer) prior to the first dose of the study drug pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 and above National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 toxicity attributed to combination treatment | Up to 180 days post-SBRT
  The toxicity profiles will be tabulated by follow-up period (i.e. 30 days and 180 days).

SECONDARY OUTCOMES:
Response rate, assessed using RECIST | Up to 24 months
  Estimated based on the number of responses using a binomial distribution and its confidence intervals will be estimated using Wilson's method. Factors including patient characteristics that predict response will be identified by logistic regression.
Change in tumor volume | Baseline to up to 24 months
  Summarized by mean ± standard deviation and the difference between two time points (pre and post treatment) will be examined using paired T-test.
Disease-free survival | From the start of treatment to the date of disease progression or the date of death, whichever comes first, assessed up to 24 months
  Summarized by calculating Kaplan-Meier curves. Survival rates estimated from the Kaplan-Meier curves will be estimated with 95% confidence intervals.
Overall survival | From the start of treatment to the date of death, assessed up to 24 months
  Summarized by calculating Kaplan-Meier curves. Survival rates estimated from the Kaplan-Meier curves will be estimated with 95% confidence intervals.
Time to local progression | From the start of treatment to the date of local progression, assessed up to 24 months
  Summarized by calculating Kaplan-Meier curves. Survival rates estimated from the Kaplan-Meier curves will be estimated with 95% confidence intervals.
Time to distant failure | From the start of treatment to the date of distant metastases, assessed up to 24 months
  Summarized by calculating Kaplan-Meier curves. Survival rates estimated from the Kaplan-Meier curves will be estimated with 95% confidence intervals.
Rate of acute side effects | Up to 180 days after treatment
  Summarized as a proportion with 95% confidence intervals.
Rate of late side effects | Up to 24 months
  Summarized as a proportion with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Ellis, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio